CLINICAL TRIAL: NCT06740890
Title: A Proof of Concept Study of Time Limited Exercise Plus Olanzapine-samidorphan for the Prevention of Early Weight Gain
Brief Title: Exercise and Olanzapine-samidorphan
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Joshua Kantrowitz, Associate Professor, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2028
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Schizophenia Disorder; Schizoaffective Disorder; Bipolar Disorder I or II; Bipolar Disorder NOS
Keywords: Exercise; Antipsychotic induced weight gain; olanzapine-samidorphan
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- olanzapine-samidorphan plus exercise (Experimental)
  Interventions: Drug: Olanzapine-samidorphan + exercise

INTERVENTIONS:
Drug: Olanzapine-samidorphan + exercise — 8 weeks of open label Olanzapine-samidorphan + 4 weeks of aerobic exercise

SUMMARY:
This is a single site trial in 30 patients with schizophrenia, schizoaffective, or bipolar I/II/NOS disorder in which all participants will receive eight weeks of olanzapine and samidorphan (Olz/Sam) plus four weeks of aerobic exercise.

DETAILED DESCRIPTION:
The principal hypothesis is that Olz/Sam combined with aerobic exercise will lead to less weight gain than Olz/Sam alone (historical data) when measured at 4 weeks. People with schizophrenia, schizoaffective and bipolar disorder I,II and NOS are eligible.

After informed consent, patients will undergo a full medical/psychiatric screening and be assessed for a reason to switch antipsychotic medication. Eligible subjects will receive 8 weeks of open label Olz/Sam. Over the first 4 weeks of treatment, all subjects will complete 4 weeks of aerobic exercise for 2 to 4 days a week. Olanzapine will be flexibly dosed over the first 4 weeks according to investigator discretion. The Sam dose will remain fixed at 10 mg for the duration of the study.

Subjects will undergo comprehensive weight, metabolic, and symptomatic assessments before and after 4 weeks of exercise, and again at study end (8 weeks). Cognitive assessments will be done at Visit 2/Baseline and study end.

This is a single site study.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65, inclusive at Visit 1.
2. DSM-V diagnosis of schizophrenia or schizoaffective or Bipolar I/II/NOS disorder at Visit 1.
3. Body Mass Index (BMI) of 18.0-40.0 kg/m2, inclusive, at Visits 1 and 2.
4. Willing to provide informed consent at Visit 1.
5. Medically and psychiatrically stable for study participation at Visit 1.
6. Responsive to an antipsychotic treatment (other than clozapine) in the past 5 years prior to Visit 1.
7. Can benefit from participation in this study and has a reason to participate, such as inadequate efficacy on current treatment, side effects on current treatment, desire to start olanzapine-samidorphan or try structured exercise program (assessed at Visit 1).
8. Maintained a stable body weight (change < 5%) for at least 3 months prior to Visit 1.
9. Willing to use qualified methods of contraception (listed in section 5.3) for the study duration (for women of childbearing potential only) (assessed at Visit 1 and Visit 2).

Exclusion Criteria:

1. Positive drug screen for opioids, phencyclidine, amphetamine/ methamphetamine, or cocaine at Visit 1 or Visit 2.
2. Diagnosis of moderate or severe substance use disorder, anorexia nervosa, bulimia, binge eating disorder or any other clinically significant eating disorder at Visit 1.
3. EKG abnormality that is clinically significant including a QT interval > 450 msec for men and > 470 msec for women, as corrected by the Fridericia formula (QTcF) at Visit 1.
4. Use of olanzapine+samidorphan for any reason in the last six months prior to Visit 1, any history of poor or inadequate response to treatment with olanzapine or no justifiable reason to expect improvement on olanzapine as assessed at Visit 1.
5. Taken opioid agonists (e.g., codeine, oxycodone, tramadol, or morphine) within the 14 days prior to Visit 1 and/or anticipates a need to take opioid medication during the study period (e.g., planned surgery), or has taken opioid antagonists including naltrexone (any formulations) or naloxone within 60 days prior to Visit 1.
6. Pregnant or breast feeding women. Women of child-bearing potential must have a negative serum beta-hCG pregnancy test at Visit 1 and a negative urine pregnancy test at Visit 2.
7. Any clinically significant or unstable medical illness, condition, or disorder that is anticipated to potentially compromise subject safety on study medication or exercise, or adversely affect the evaluation of efficacy, including (but not necessarily limited to) the following (as assessed at Visit 1):

   1. Clinically significant hypotension or hypertension not stabilized on medical therapy.
   2. Unstable thyroid dysfunction in the past 6 months (e.g., hypothyroidism, hyperthyroidism, or thyroiditis that was untreated, or discovered and treatment was initiated within the 6 months prior to screening).
   3. Personal or family history of neuroleptic malignant syndrome, has a history of clinically significant extrapyramidal symptoms when taking olanzapine, or has had clinically significant tardive dyskinesia.
   4. Neurological conditions include the following:

      * History of seizure disorder or a condition associated with seizures (except history of febrile seizures).
      * History of brain tumor, subdural hematoma, stroke or any other clinically significant neurological condition within the 12 months prior to Visit 1.
      * Head trauma with loss of consciousness within the 12 months prior to Visit 1.
      * Active, acute or chronic CNS infection.
   5. Cardiac condition that might confound study results, pose additional risk when administering the study drug or exercise regimen to the subject, or preclude successful completion of the study. Conditions include the following:

      * Clinically significant cardiac arrhythmia, cardiomyopathy, a cardiac conduction defect, or a history of myocardial infarction or unstable angina within 6 months prior to Visit 1.
8. Currently taking any contraindicated medications as per the approved labeling for Olz-Sam (see section 6.5 for details) at Visit 1 and Visit 2.
9. Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 3 months prior to Visit 1 or current at Visit 2
10. Inflammatory bowel disease or any other gastrointestinal disorder associated with weight loss at Visit 1.
11. Joined a weight management program or had significant changes in diet or exercise regimen within 6 weeks prior to Visit 1 or plans to join a weight management program during the study as assessed at Visit 1.
12. History of diabetes (assessed at Visit 1).
13. Laboratory abnormality that would compromise the well-being of the subject, or any of the following specific laboratory results at Visit 1:

    1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value > 2 times the upper limit of the laboratory normal reference range
    2. Absolute neutrophil count (ANC) <1.5 x 10^3 μL
    3. Platelet count < 75 x 10^3 uL
    4. Serum creatinine > 1.5 mg/dL
    5. Dyslipidemia, defined for this study as total fasting cholesterol > 280 mg/dL or fasting triglycerides > 500 mg/dL
    6. Hemoglobin A1c (HbA1c) > 6.0%
    7. Fasting plasma glucose > 126 mg/dL (7.0 mmol/L)
14. Is not fit for the trial in the opinion of the investigator at Visit 1 and Visit 2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Weight | 4 weeks
  Body weight

SECONDARY OUTCOMES:
Weight | 8 weeks
  4 weeks post formal exercise program

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
non-PHI upon request
Supporting Information: Study Protocol, ICF
Time Frame: six months after publication
Access Criteria: upon request

REFERENCES:
- [Background] Huhn M, Nikolakopoulou A, Schneider-Thoma J, Krause M, Samara M, Peter N, Arndt T, Backers L, Rothe P, Cipriani A, Davis J, Salanti G, Leucht S. Comparative efficacy and tolerability of 32 oral antipsychotics for the acute treatment of adults with multi-episode schizophrenia: a systematic review and network meta-analysis. Lancet. 2019 Sep 14;394(10202):939-951. doi: 10.1016/S0140-6736(19)31135-3. Epub 2019 Jul 11. PMID 31303314
- [Background] Correll CU, Newcomer JW, Silverman B, DiPetrillo L, Graham C, Jiang Y, Du Y, Simmons A, Hopkinson C, McDonnell D, Kahn RS. Effects of Olanzapine Combined With Samidorphan on Weight Gain in Schizophrenia: A 24-Week Phase 3 Study. Am J Psychiatry. 2020 Dec 1;177(12):1168-1178. doi: 10.1176/appi.ajp.2020.19121279. Epub 2020 Aug 14. PMID 32791894